CLINICAL TRIAL: NCT01478841
Title: INFLUENCE OF POLYPHENOLS ON OXIDATIVE STRESS IN HEALTHY INDIVIDUALS WITH HIGH METABOLISM RISK: RELATIONSHIP WITH THE MECHANISMS OF INSULIN RESISTANCE
Brief Title: Polyphenols and Insulin Resistance
Acronym: POLYOXRESIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UF8178
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Healthy Volunteers; Insulin Resistance; Type 2 Diabetes (T2D)
Keywords: insulin resistance; type 2 diabetes (T2D); cardiovascular complications; polyphenolic compounds derived from red grape marc extracts; oxidative stress
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Polyphenols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polyphenols (Experimental): 9 weeks of supplementation with polyphenols(D56) and during the last week supplementation with polyphenols associated with a fructose load during the last 6 days (D63).
  Interventions: Drug: polyphenol
- placebo (Placebo Comparator): 9 weeks of supplementation with placebo (D56) and during the last week supplementation with placebo associated with a fructose load during the last 6 days (D63).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: polyphenol — 2 capsules of 0.5 gram to be taken at the beginning of breakfast and dinner (2g/day) fructose : dose of 3 g/kg/day from D57 to D62 in the form of a 20% solution taken during the three main meals
  Arms: Polyphenols
Drug: placebo — 2 capsules of 0.5 gram to be taken at the beginning of breakfast and dinner (2g/day) fructose : dose of 3 g/kg/day from D57 to D62 in the form of a 20% solution taken during the three main meals
  Arms: placebo

SUMMARY:
Diet and nutrition play an essential role in the development and the clinical expression of the most common health problems. Overeating and obesity induce oxidative stress, which has been proposed to be a pathogenic mechanism leading to insulin resistance, type 2 diabetes (T2D) and associated cardiovascular complications. The main objective of the proposed research is to evaluate the beneficial effects of polyphenolic compounds derived from red grape marc extracts on the cascade of events leading from overeating to oxidative stress and insulin resistance. For that, we will study free radicals production, inflammatory markers, adipokines, mitochondrial function, insulin sensitivity and energy substrate utilization in healthy volunteers at risk for insulin resistance and T2D (1st degree relatives of T2D patients with associated overweight). These volunteers will be randomized between a placebo and a polyphenol group for 9 weeks. The demonstration of the beneficial effects of polyphenols will be sensitized by high-fructose feeding for the last 6 days of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Absence of anti HIV or anti hepatitis C antibodies and of HBS antigen.
* Acceptable biological assessment of the hepatic and renal functions (γGT, ALAT, ASAT < 3 times the normal value and serum creatinine <150 micromol/l).
* Age between 30 and 55 years.
* Fasting plasma glucose <110 mg/dl and absence of any anti-diabetic treatment
* No regular physical activity (Voorips index < 9)
* Absence of any drug treatment in progress and during the last 2 months
* Subjects with at least one 1st degree relative with T2D and with a body mass index between 25 and 35 kg/m² and a waist measurement >94 cm for males, and >80 cm for females.
* Normal ionogram (sodium 135 - 145 mmol/l, potassium 3,5 - 4,5 mmol/l).
* Normal ferritin level (75 - 300 ng/ml)
* hs-CRP <8 mg/l.
* Absence of arterial hypertension (systolic pressure <140 mmHg and diastolic pressure <90 mmHg).
* Non smoker or former smoker (quit smoking >1 year).
* Alcohol consumption <30 g/day.

Exclusion Criteria:

* Hyperthermia (T°>38°c)
* Subject deprived of freedom by a court or administrative order
* Major protected by the law
* Subject who is in a period of relative exclusion due to his/her participation to another protocol or for whom the annual maximum amount of allowances of 3 811.23 € is reached.
* Subject who has been treated with anti-coagulants, anti-inflammatory drugs, b-blockers or insulin during the last month.
* Subject who cannot be subjected to muscle biopsy.
* Allergy to the anaesthetic
* Woman in age to procreate and not taking any oral or intra-uterine contraception

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Peripheral insulin-sensitivity | 6 weeks

SECONDARY OUTCOMES:
biochemical parameters | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France

REFERENCES:
- [Derived] Hokayem M, Blond E, Vidal H, Lambert K, Meugnier E, Feillet-Coudray C, Coudray C, Pesenti S, Luyton C, Lambert-Porcheron S, Sauvinet V, Fedou C, Brun JF, Rieusset J, Bisbal C, Sultan A, Mercier J, Goudable J, Dupuy AM, Cristol JP, Laville M, Avignon A. Grape polyphenols prevent fructose-induced oxidative stress and insulin resistance in first-degree relatives of type 2 diabetic patients. Diabetes Care. 2013 Jun;36(6):1454-61. doi: 10.2337/dc12-1652. Epub 2012 Dec 28. PMID 23275372